CLINICAL TRIAL: NCT07316816
Title: Stanford Pediatric Healthy Weight Index
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Karl Sylvester, Professor of Surgery, Stanford University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 81022
Record Dates: First submitted 2025-12-08; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Obesity & Overweight
Keywords: Metabolism; Continuous Glucose Monitoring; Obesity; Bariatric Surgery; GLP-1
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Bariatric Surgery (Experimental): Adolescent patients in the Adolescent Bariatric Program at Stanford Children's undergoing bariatric surgery will undergo continuous glucose monitoring and fitness tracking throughout the course of study.
  Interventions: Other: Remote Monitoring Program
- GLP-1 (Experimental): Adolescent patients being considered for GLP-1 receptor agonist therapy for obesity management will undergo continuous glucose monitoring and fitness tracking throughout the course of study.
  Interventions: Other: Remote Monitoring Program

INTERVENTIONS:
Other: Remote Monitoring Program — Continuous glucose monitors will be placed at 2 or 3 clinically relevant time points and participants will track their fitness using wearable devices.

SUMMARY:
This study will develop a simple index to measure how well the body uses insulin and overall heart and metabolic health in children and teens with obesity. The investigators will use data from wearable devices (like fitness trackers) and glucose monitors, along with lab tests, to learn how activity and glucose relate to metabolic problems.

DETAILED DESCRIPTION:
This is a prospective cohort study to develop a metabolic index for insulin sensitivity and cardiometabolic fitness among children and adolescents with obesity. Adolescent patients undergoing evaluation for bariatric surgery or medical management of wight using GLP-1 agonist therapies will be consented for participation. Participants will be given a wearable fitness device and a continuous glucose monitor. Continuous monitoring will be carried out at three time points: preoperative or prior to starting medication, perioperative or after 3-4 weeks of GLP1 use during early treatment phase, and 3 months post-operatively or 3 months after dose stabilization or discontinuation.

ELIGIBILITY:
Inclusion Criteria:

* Class 2 and 3 obesity
* Patient in the Adolescent Bariatric Program at Stanford Children's that is eligible for either laparoscopic sleeve gastrectomy or GLP1 Receptor Agonist Therapy
* Willingness to wear a CGM and physiological monitor for the duration of the study.

Exclusion Criteria:

* Hypothalamic and syndromic obesity
* BMI > 55
* Plan to undergo bariatric surgical procedure other than sleeve gastrectomy
* Prior bariatric surgical procedure
* Active GLP treatment (within past 3 months)
* Unable to read, understand, or complete the informed consent in English or Spanish

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-01-05 (Estimated); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Percent Reduction in BMI | baseline through study completion, an average of 4 months
  assessment of change in BMI from pre-intervention to post-intervention
Body Weight | baseline through study completion, an average of 4 months
  Change in body weight (kg)
Fasting Glucose | baseline through study completion, an average of 4 months
  change in fasting glucose levels from pre-intervention to post-intervention
Fasting Insulin | baseline through study completion, an average of 4 months
  change in fasting insulin levels from pre-intervention to post-intervention
HbA1c | baseline through study completion, an average of 4 months
  change in HbA1c levels from pre-intervention to post-intervention
Lipid Panel | baseline through study completion, an average of 4 months
  changes in lipid panel levels from pre-intervention to post-intervention
Liver Enzymes | baseline through study completion, an average of 4 months
  changes in liver enzymes from pre-intervention to post-intervention

SECONDARY OUTCOMES:
Obesity-related Comorbidities | baseline through study completion, an average of 4 months
  Defined as resolution or improvement according to prespecified clinical criteria

CONTACTS AND LOCATIONS:
Locations (1):
- Lucile Packard Children's Hospital - Stanford, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No